CLINICAL TRIAL: NCT06280937
Title: Short Term Effect of Wearing a Tie on Musculoskeletal System
Brief Title: Short Term Effect of Wearing a Tie
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Omer Dursun, Asst. Prof., Bitlis Eren University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BEUFTR-2
Record Dates: First submitted 2024-02-15; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Musculoskeletal Disorder
Keywords: spine; pain threshold
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Control group will go on their routine daily activities. Study group will wear a tie during one office working day.
Who Masked: Outcomes Assessor
Masking Description: Interventions and assessment will be performed by separate researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): In this group, participants will go on their daily activities. No additional intervention will be applied to the participants in this group.
- Study Group (Experimental): In this group, participants will wear a tie during one office working day
  Interventions: Other: Wearing a tie

INTERVENTIONS:
Other: Wearing a tie — Individuals in the study group will be asked to wear a tie during one office working day.
  Arms: Study Group

SUMMARY:
The goal of this randomized controlled study is to assess the short term effect of wearing a ties on musculoskeletal system. In this scope viscoelastic properties and the mechanosensitivity of the muscles, and cervical range of motion will be measured. In addition to these measurements activity limitation due to wearing a tie and trunk mobility will be assessed.

DETAILED DESCRIPTION:
A total of at least 54 volunteers who satisfies the eligibility criteria of the study will be recruited to the study. Following to the recruitment process participants will be randomly assigned to the one of the two groups. Participants in the control group will go on to their daily activities. Participants in the study group will be asked to wear a tie for one working day.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 25 years
* Given a signed consent
* Low level of physical activity
* Having a BMI between 18 kg/m2 and 25 kg/m2
* No pain in neck, upper and lower back (numerical pain rating scale below 3 points)

Exclusion Criteria:

* Having a systemic or metabolic disease
* Having a mental disorder
* Chronic drug use
* Any condition that may result in muscle atrophy
* Musculoskeletal surgery history in last 3 months
* Having a cervical, thoracal or lumbar radiculopathy or myelopathy
* Having a whiplash syndrome or fibromyalgia
* Having performed any strenuous exercises within the 24 h prior to measurements

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants' gender must be stated as male in their identity
Enrollment: 54 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
The Change in the Viscoelastic Properties of the Muscles | Change from baseline pain at eight hours and one day
  The effect of wearing a tie on the viscoelastic properties of participants' upper trapezius, cervical, thoracic, and lumbar paravertebral muscles will be measured using the myotonometer (MyotonPRO). Tonus measurement of the trapezius muscle will be taken from the upper, middle and lower part of the muscle. Evaluation of cervical muscle tone will be conducted 2 cm to the right and left of the C4 spinous process. The measurement will be taken on the semispinalis capitis muscle while the individual lies face down on the treatment bed. Muscle tone measurements for the thoracic and lumbar regions will be taken on the paravertebral muscles at the T3, T7, T11, L1 and L4 levels.
The Change in the Pressure Pain Threshold of the Spine and Upper Trapezius | Change from baseline mechanosensitivity at eight hours and one day
  The potential impact of wearing a tie on individuals' pain thresholds will be evaluated using an analog algometer. Pain threshold measurements will be taken at the upper trapezius muscle, C6, T6, and L4 vertebral spinous processes. The algometer will be positioned perpendicular to the measurement areas. Three measurements will be taken for each region, with a half-minute interval between measurements. The average of the three measurements will be calculated and recorded. A change of 20-25% in the algometric measurement values will be considered significant.
Cervical Range of Motion | Change from baseline cervical range of motion at immediate, eight hours and one day
  The effect of wearing a tie on participants' cervical range of motion will be measured using a 10-inch standard manual goniometer. For measuring cervical flexion and extension range of motion, the pivot point of the goniometer will be placed at the external auditory meatus. The fixed arm of the goniometer will be held vertically, and the moving arm will follow along the base of the nostrils. To measure cervical rotation range of motion, measurements will be taken from behind the participants. The pivot point of the goniometer will be placed at the vertex, while the fixed arm will be kept parallel to the acromion and the moving arm will follow along with their nose. Lateral flexion range of motion will be taken in front of the participants. The pivot point of the goniometer will be placed over the sternal notch, with its fixed arm parallel to the acromion and its moving arm will follow along tip of the participants' nose. Each range of motion measurement will be performed three times.

SECONDARY OUTCOMES:
Activity Limitation | Change from baseline activity limitation at eight hours
  The activities that individuals find difficult due to wearing a tie will be assessed using a visual analog scale. Individuals will be asked to rate three activities they find difficult while wearing a tie on a scale from 0 to 10. A score of 0 indicates no difficulty, while a score of 10 indicates that performing the activity is nearly impossible.
Global Rating of Change | Change from baseline global rating of change at eight hours
  In the study group, the Global Rating of Change Scale (GROC) will be used to assess the changes experienced by individuals after wearing a tie. The scale ranges from "-7" to "+7" and consists of a total of 15 points. A score of "-7" indicates a much worse condition, while a score of "+7" indicates a much better condition.
Trunk Forward Bending Mobility | Change from baseline cervical range of motion at immediate, eight hours and one day
  The potential effect of wearing a tie on trunk flexion mobility will be assessed using the fingertip-to-floor test. In the fingertip-to-floor test, individuals will be asked to stand barefoot and adjacent to a platform of 20 cm in height without bending their knees, toes, or arms, and to lean forward towards their toes. Then, the distance from the ground will be measured using a measuring tape. The measurement will be repeated twice, and the average of the measurements will be taken.
Trunk Lateral Bending Mobility | Change from baseline cervical range of motion at immediate, eight hours and one day
  The potential effect of wearing a tie on trunk lateral bending mobility will be assessed using the fingertip-to-floor test. In the fingertip-to-floor test, individuals will be asked to stand barefoot and adjacent to a platform of 20 cm in height without bending their knees, toes, or arms, and to bend laterally towards their toes. Then, the distance from the ground to the tip of the middle finger will be measured using a measuring tape. The measurement will be repeated twice, and the average of the measurements will be taken.
Neck Circumference | At baseline
  While the participant looking straight ahead, with relaxed shoulders (not hunched), middle and lower neck circumference will be measured with the measuring tape.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Dursun, Asst. Prof., Principal Investigator — Bitlis Eren University; Erhan Dincer, M.Sc., Principal Investigator — Bitlis Eren University; Cihan Önen, Asst. Prof., Principal Investigator — Bitlis Eren University; Deniz Akbulut, M.D., Principal Investigator — Van Training and Research Hospital
Locations (1):
- Bitlis Eren University, Bitlis, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoo IG, Kim MH, Yoo WG. Effects of wearing a tight necktie on cervical range of motion and upper trapezius muscle activity during computer work. Work. 2011;39(3):261-6. doi: 10.3233/WOR-2011-1174. PMID 21709362
- [Background] Usgu S, Ramazanoglu E, Yakut Y. The Relation of Body Mass Index to Muscular Viscoelastic Properties in Normal and Overweight Individuals. Medicina (Kaunas). 2021 Sep 26;57(10):1022. doi: 10.3390/medicina57101022. PMID 34684059
- [Background] Ramazanoglu E, Turhan B, Usgu S. Evaluation of the tone and viscoelastic properties of the masseter muscle in the supine position, and its relation to age and gender. Dent Med Probl. 2021 Apr-Jun;58(2):155-161. doi: 10.17219/dmp/132241. PMID 34076970
- [Background] Wu Z, Zhu Y, Xu W, Liang J, Guan Y, Xu X. Analysis of Biomechanical Properties of the Lumbar Extensor Myofascia in Elderly Patients with Chronic Low Back Pain and That in Healthy People. Biomed Res Int. 2020 Feb 18;2020:7649157. doi: 10.1155/2020/7649157. eCollection 2020. PMID 32149135
- [Background] Tawde P, Dabadghav R, Bedekar N, Shyam A, Sancheti P. Assessment of cervical range of motion, cervical core strength and scapular dyskinesia in violin players. Int J Occup Saf Ergon. 2016 Dec;22(4):572-576. doi: 10.1080/10803548.2016.1181892. Epub 2016 May 27. PMID 27232160
- [Background] Youdas JW, Carey JR, Garrett TR. Reliability of measurements of cervical spine range of motion--comparison of three methods. Phys Ther. 1991 Feb;71(2):98-104; discussion 105-6. doi: 10.1093/ptj/71.2.98. PMID 1989013
- [Background] Ylinen J, Takala EP, Kautiainen H, Nykanen M, Hakkinen A, Pohjolainen T, Karppi SL, Airaksinen O. Effect of long-term neck muscle training on pressure pain threshold: a randomized controlled trial. Eur J Pain. 2005 Dec;9(6):673-81. doi: 10.1016/j.ejpain.2005.01.001. PMID 16246820
- [Background] Ruiz-Saez M, Fernandez-de-las-Penas C, Blanco CR, Martinez-Segura R, Garcia-Leon R. Changes in pressure pain sensitivity in latent myofascial trigger points in the upper trapezius muscle after a cervical spine manipulation in pain-free subjects. J Manipulative Physiol Ther. 2007 Oct;30(8):578-83. doi: 10.1016/j.jmpt.2007.07.014. PMID 17996549
- [Background] Sanchez-Infante J, Bravo-Sanchez A, Jimenez F, Abian-Vicen J. Effects of dry needling on mechanical and contractile properties of the upper trapezius with latent myofascial trigger points: A randomized controlled trial. Musculoskelet Sci Pract. 2021 Dec;56:102456. doi: 10.1016/j.msksp.2021.102456. Epub 2021 Sep 3. PMID 34507046
- [Background] Liu CL, Feng YN, Zhang HQ, Li YP, Zhu Y, Zhang ZJ. Assessing the viscoelastic properties of upper trapezius muscle: Intra- and inter-tester reliability and the effect of shoulder elevation. J Electromyogr Kinesiol. 2018 Dec;43:226-229. doi: 10.1016/j.jelekin.2017.09.007. Epub 2017 Oct 19. PMID 29103836